CLINICAL TRIAL: NCT05975801
Title: Investigation of the Effectiveness of Dry Cupping Therapy on Rotator Cuff Injuries
Brief Title: Dry Cupping Therapy on Rotator Cuff Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sumeyye tunc, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMU-FTR-ST-02
Record Dates: First submitted 2023-07-25; First posted 2023-08-04 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Injuries; Shoulder Pain; Subacromial Impingement Syndrome
Keywords: Complementary Therapies; Cupping Therapy; Range of Motion; Rotator Cuff Injuries; Shoulder Pain; Quality of Life
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Shoulder Impingement Syndrome | interventions — Conservative Treatment; Transcutaneous Electric Nerve Stimulation; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Cupping Therapy Group (Active Comparator): In addition to the conventional treatment, moving cup application was applied for 10 minutes twice a week. During the treatment, the patients were placed in a side-lying position with the affected side on top. Liquid petroleum jelly was applied on the skin and negative pressure was created with a manual pump, allowing the cup to be slid on the skin. Care was taken to ensure that the negative pressure would not cause increased pain and would allow the cup to slide. Deltoid, Trapeze, Supraspinatus, Infraspinatus, Pectoral muscles were applied in the origo insertion direction for a total of 10 minutes.
  Interventions: Other: Dry Cupping Therapy; Other: Conservative Treatment (hotpack, transcutaneous electrical nerve stimulation(TENS), ultrasound
- Conservative Treatment Group (Other): The patients in the control group received a conservative treatment program including hotpack (20 min), transcutaneous electrical nerve stimulation(TENS) (COMPEX Rehab 400 - 20 min), ultrasound (Chattanooga Ultrasound - 1 megahertz, 1.5 W/cm², 5 min) for 4 weeks, 5 days a week, and wand, Codman, stretching and strengthening exercises were applied.Stretching exercises were added to the treatment for the shoulder girdle and scapular region muscles, while strengthening exercises were added to the treatment by increasing the resistance at the pain limit. In addition, the home exercise program was taught to be 10 repetitions 2 times a day.
  Interventions: Other: Conservative Treatment (hotpack, transcutaneous electrical nerve stimulation(TENS), ultrasound

INTERVENTIONS:
Other: Dry Cupping Therapy
  Arms: Dry Cupping Therapy Group
Other: Conservative Treatment (hotpack, transcutaneous electrical nerve stimulation(TENS), ultrasound

SUMMARY:
Shoulder pain is the most common musculoskeletal problem after spine and knee complaints. Rotator cuff injuries (RCI) are the most common cause of shoulder pain. RCI includes a wide spectrum from subacromial impingement syndrome (SIS) to chronic tendinopathy, partial and total ruptures of the rotator cuff. In recent years there has been a renewed interest in traditional and complementary medicine (TCM) for various musculoskeletal problems. Cupping therapy, which is one of the most commonly used TCM methods, is one of the oldest medical applications with thousands of years of history. Although it is thought to be effective in many diseases, there are not enough studies in the literature about its effectiveness and mechanism of action. Our aim in this study is to investigate the effects of moving dry cupping therapy on pain, range of motion (ROM), functionality and quality of life in RCI.

DETAILED DESCRIPTION:
Shoulder pain is the most common musculoskeletal problem after spine and knee complaints. Rotator cuff injuries (RCI) are the most common cause of shoulder pain. RCI includes a wide spectrum from subacromial impingement syndrome (SIS) to chronic tendinopathy, partial and total ruptures of the rotator cuff. Conservative and surgical techniques are used in the treatment. Conservative treatments; various medical treatments, activity modifications, hot and cold agents, exercise, manual therapy, acupuncture, electrophysical agents, etc. includes applications. In recent years there has been a renewed interest in traditional and complementary medicine (TCM) for various musculoskeletal problems. Cupping therapy is an ancient TCM treatment that has been practiced in different ways in many cultures in Asia, Europe and the Middle East throughout history, but its true origin remains unclear. Although cupping therapy has been used to treat pain and various complaints for thousands of years, it has almost disappeared from the therapeutic spectrum of Western medicine with pharmacological developments in the late 20th century. However, over the past few years, interest in the cup has increased, and new clinical research suggests that the cup may be potentially effective in the management of painful conditions, in the treatment of pain-related diseases. Although it is stated in the literature that it is used in the treatment of many neuromusculoskeletal problems, according to the information participants have obtained in the relevant literature, there is not yet a study examining the effects of cupping therapy in RCI. In the light of these data, our aim in this study is to investigate the effects of moving dry cupping therapy on pain, range of motion (ROM), functionality and quality of life in RCI.Hypotheses:

H0: Cupping therapy has no effect on improving pain, ROM, functionality and quality of life in individuals with RCI.

H1: Cupping therapy has an effect on improving pain, ROM, functionality and quality of life in individuals with RCI.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 age range
* Clinical diagnosis ofRCI, SIS, supraspinatus tendinitis
* To be fully cooperative

Exclusion Criteria:

* Patients who had undergone any surgical operation on the shoulder
* A history of shoulder fracture
* Severe osteoporosis
* Total tendon rupture
* Had received oral/intramuscular steroids in the last 1 month
* Had been administered intra-articular drugs in the last 3 months
* Difficulty in cooperation

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain | 1 months
  Pain was evaluated with the Numerical Rating Scale (NRS). The patient was asked to mark his pain in numerical values ranging from 0 (no pain) to 10 (very severe pain). The higher the score obtained from this test, the more pain the patient has, and the smaller the score, the less the pain is predicted.
Range of Motion | 1 months
  Shoulder flexion, abduction, internal and external rotation in the supine position using a baseline goniometer; Shoulder extension ROM in the prone position was evaluated as passive.
Constant-Murley Score | 1 months
  Developed in 1987, this scoring system evaluates pain, activities of daily living, strength, and ROM. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively. In the original publication, the pain experienced during normal activities of daily living was scored as: no pain = 15 points, mild = 10, moderate = 5 and severe = 0 points
The Disabilities of the Arm, Shoulder and Hand (DASH) | 1 months
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100
Short Form (SF-36) | 1 months
  SF-36, which is one of the most preferred scales in assessing the quality of life, consists of a total of 36 questions and 8 sections. It is divided into 8 parts as physical function, social function, physical role difficulty, emotional role difficulty, mental health, energy/vitality, pain and general health perception. Each section is scored between 0-100 in itself. High scores indicate high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Esra ATILGAN, Study Director — Medipol University; Hatice Hümeyra AKIL, Principal Investigator — Uskudar University; Sümeyye TUNÇ, Study Chair — Medipol University